CLINICAL TRIAL: NCT07096960
Title: A Brazilian Version of the STrAtegies for RelaTives (START) Intervention in the Unified Health System (SUS): a Controlled Feasibility Trial
Brief Title: Implementation of the START Intervention in Brazil: a Controlled Feasibility Trial
Acronym: START/ESCADA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Alemão Oswaldo Cruz (Other)
Collaborators: University College, London (Other); Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Lucas Martins Teixeira, Principal Investigator, Hospital Alemão Oswaldo Cruz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PC CEP HAOC 7.432.280
Record Dates: First submitted 2025-06-25; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Caregiver Burden of People With Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- START/ESCADA Intervention (Experimental): Participants will receive the culturally adapted Brazilian version of START (ESCADA).
  Interventions: Behavioral: STrAtegies for RelaTives (START) - Brazilian version
- Waitlist Control (No Intervention): Participants receive usual care and will be offered the START/ESCADA intervention after 6 months at the end of the study.

INTERVENTIONS:
Behavioral: STrAtegies for RelaTives (START) - Brazilian version — Eight individualized, weekly, home-based sessions will be delivered by trained community general health workers (CGHW). The intervention includes coping strategies, behavior management, and communication skills. Caregivers receive printed materials and structured exercises. CGHW receive a facilitator manual.
  Arms: START/ESCADA Intervention

SUMMARY:
This controlled trial aims to assess the feasibility of a culturally adapted Brazilian version of the START (STrAtegies for RelaTives) program, a structured coping strategy program designed for family caregivers of people living with dementia. The program will be delivered by trained community general health workers (CGHW) in 10 municipalities across Brazil. Outcomes will include measures of feasibility and acceptability, as well as caregiver burden, mental health, and quality of life, assessed at baseline and after 6 months.

DETAILED DESCRIPTION:
This study will evaluate the feasibility of the START program in the Brazilian Unified Health System (SUS). The intervention was translated and culturally adapted through a structured process that included expert review and focus groups with mental health professionals and community general health workers (CGHW) to ensure the clarity and cultural relevance of the materials.

The intervention will be delivered by trained CGHW to family caregivers of people living with dementia. CGHW will undergo a 16-hour, in-person training provided by the research team. During the period of the intervention, they will receive ongoing remote supervision to support protocol adherence and address challenges encountered in the field.

Ten municipalities-two from each of the five geographical regions of Brazil-will participate. In each municipality, two primary care units (PCU) will be randomly allocated to either the intervention or the waitlist control group.

The selection of participating municipalities will be conducted in collaboration with each state's Bipartite Inter-managerial Commission (Comissão Intergestora Bipartite, CIB). Municipalities will be eligible if they have ≥100,000 inhabitants and agree to participate. Each will be required to list all PCU with ≥15 dementia diagnoses (ICD-10). If a municipality does not have at least two PCU meeting this threshold, units with ≥10 diagnoses may be considered. From this list, two PCU will be randomly drawn. Eligible pairs must meet two conditions: (1) they must be non-contiguous, and (2) their populations must be demographically similar, as assessed by local authorities. If these two criteria are not met, a new draw will be conducted.

Feasibility and acceptability will be assessed as primary outcomes through operational indicators (e.g., number of sessions completed, adherence, dropouts), structured online questionnaires completed by caregivers and CGHW, and semi-structured qualitative interviews conducted with caregivers, CGHW, and municipal health managers.

Secondary outcomes will include caregiver burden, mental health symptoms, quality of life, coping strategies, and neuropsychiatric symptoms of the care recipient. These outcomes will be measured at baseline and again six months after the intervention using validated instruments including the HADS, ZBI, WHOQOL-Bref, Brief COPE, and NPI.

Intervention fidelity will be assessed through randomly selected audio recordings of sessions and structured checklists completed by independent researchers.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregivers (≥18 years old) who are the primary or one of the primary persons responsible for caring for a family member with dementia, providing regular and sustained emotional or practical support every week, and living in the same household or nearby with frequent face-to-face interaction.
* Care recipient (person with dementia) with Clinical Dementia Rating (CDR) score ≥1.
* Care recipient with at least one ICD-10 dementia diagnosis code documented in their medical record.

Exclusion criteria:

* Illiterate caregivers.
* Caregivers who provide only occasional or sporadic support (less than weekly or without regular caregiving responsibility).
* Care recipients who are institutionalized (e.g., living in long-term care facilities).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility questionnaire | Approximately 8 weeks post-baseline (after completing the intervention)
  Feasibility of the START/ESCADA intervention assessed through an online structured questionnaire applied to caregivers and community health workers (CHW), covering domains of acceptability, demand, implementation, practicality, adaptation, integration, and expansion.
Operational feasibility metrics | Approximately 8 weeks post-baseline (after completing the intervention)
  Number of caregivers who consented to participate; number and proportion who completed all 8 sessions; average number of weeks to complete 8 sessions; number and proportion of community health workers (CHW) completing training; number of CHW delivering the intervention.
Qualitative feasibility interviews | Approximately 8 weeks post-baseline (after completing the intervention)
  Feasibility and acceptability of the START/ESCADA intervention assessed via semi-structured qualitative interviews with managers of primary care units, general health workers (ACS), and caregivers, exploring domains such as acceptability, demand, implementation, practicality, adaptation, integration, and expansion.

SECONDARY OUTCOMES:
Caregiver burden | 6 months post-baseline
  Zarit Burden Interview (ZBI), 22-item version; total score ranges from 0 to 88, with higher scores indicating greater caregiver burden.
Anxiety and depression | 6 months post-baseline
  Hospital Anxiety and Depression Scale (HADS); two subscales (Anxiety, Depression), each ranging from 0 to 21; higher scores indicate greater anxiety or depressive symptoms.
Quality of life (caregiver) | 6 months post-baseline
  World Health Organization Quality of Life Instrument - Short Form (WHOQOL-BREF); includes four domain scores (Physical Health, Psychological, Social Relationships, Environment), each transformed to a scale from 0 to 100; higher scores indicate better quality of life.
Coping strategies | 6 months post-baseline
  Brief COPE Inventory; 28 items grouped into 14 subscales (coping strategies), each subscale scored by summing two items (range 2 to 8); higher scores indicate greater use of the specific coping strategy.
Neuropsychiatric symptoms | 6 months post-baseline
  Neuropsychiatric Inventory (NPI); assesses 12 neuropsychiatric domains in dementia patients. Each domain score is calculated by multiplying frequency (1-4) by severity (1-3), with domain scores ranging from 0 to 12. The total NPI score ranges from 0 to 144, with higher scores indicating greater neuropsychiatric symptom burden.
Use of health and social care resources | 6 months post-baseline
  Structured questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Lucas Martins Teixeira, Vitória, Espírito Santo, Brazil